CLINICAL TRIAL: NCT01699100
Title: Reduction of Plantar Pressure in Neuropathic Diabetic Foot Patients Using Offloading Technique: Insoles With Peg Assist Design
Brief Title: Reduction of Plantar Pressure in Neuropathic Diabetic Foot Patients Using Insoles With Removable Pegs Design
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Taichung Veterans General Hospital (Other)
Responsible Party: Principal Investigator, Tung-Liang,Lin, Taichung Veterans General Hospital, Taichung Veterans General Hospital
Allocation: Not Applicable | Model: Single Group | Masking: Single | Purpose: Treatment
Other Study IDs: SF11024
Record Dates: First submitted 2012-09-26; First posted 2012-10-03 (Estimated); Last update posted 2012-10-03 (Estimated); Status verified 2012-10

CONDITIONS: Foot Ulcer, Diabetic
Keywords: offloading; plantar pressure; insole; foot ulcer
MeSH Terms: conditions — Diabetic Foot; Foot Ulcer | interventions — Equipment and Supplies

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- device (Experimental): In-shoe plantar pressure measurements were performed in 26 patients with diabetic neuropathic feet at baseline condition, and 52 regions of interest (ROIs, with mean peak pressure > 200kPa or with the highest mean peak pressure in the forefoot area) were identified as suitable areas for removal of pegs. Data of in-shoe plantar pressures of the three insole conditions (pre-peg removal, post-peg removal, and post-peg removal plus arch support) were collected. Mean peak pressure (MPP) and pressure-time integral (PTI) were recorded for analysis.
  Interventions: Other: device

INTERVENTIONS:
Other: device — Experimental: insole In-shoe plantar pressure measurements were performed in 26 patients with diabetic neuropathic feet at baseline condition, and 52 regions of interest (ROIs, with mean peak pressure > 200kPa or with the highest mean peak pressure in the forefoot area) were identified as suitable areas for removal of pegs. Data of in-shoe plantar pressures of the three insole conditions (pre-peg removal, post-peg removal, and post-peg removal plus arch support) were collected. Mean peak pressure (MPP) and pressure-time integral (PTI) were recorded for analysis.
  Other Names: Insoles from Dr.Foot Technology

SUMMARY:
The purpose of this study was to determine if insoles with removable pegs could effectively reduce the plantar aspect pressure with the aid of in-shoe plantar pressure analysis for guidance of peg removal.

DETAILED DESCRIPTION:
The investigators tested the effect of plantar pressure reduction in four conditions:

1. insole of the original shoe
2. peg assist insole but the pegs are not yet removed
3. peg assist insole and the pegs were removed
4. condition3. plus arch support to the insole

ELIGIBILITY:
Inclusion Criteria:

* previously diagnosed type 2 diabetes with neuropathic foot were recruited from the outpatient endocrinology and metabolism division of Taichung Veterans General Hospital in central Taiwan

Exclusion Criteria:

* The exclusion criteria were history of lower extremities amputation, major foot deformities, presence of active plantar foot wound or ulcer, and difficulty walking more than 100 m.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 26 (Actual)
Dates: Start 2011-09; Primary Completion 2012-05 (Actual); Study Completion 2012-05 (Actual)

PRIMARY OUTCOMES:
plantar pressure of region of interest | 30 minutes
  In-shoe plantar pressure difference between before and after insole use.

SECONDARY OUTCOMES:
Plantar pressure of non-region of interest | 30 minutes
  In-shoe plantar pressure difference between before and after insole use.

OTHER OUTCOMES:
plantar pressure of midfoot area | 30 minutes
  In-shoe plantar pressure difference between before and after insole use.

CONTACTS AND LOCATIONS:
Overall Officials: Tung-Liang Lin, MD, Principal Investigator — Taichung Verterans General Hospital

REFERENCES:
- See also: Taichung Veterans General hospital — http://www.vghtc.gov.tw/home/index.html